CLINICAL TRIAL: NCT03534310
Title: Intensive Lifestyle Modifications With or Without Liraglutide 3 mg Versus Sleeve Gastrectomy: A 3 Arm Randomized Controlled Pilot Study (LETHE)
Brief Title: Weight Loss With Intensive Lifestyle Modifications Plus Bariatric Surgery Versus Liraglutide 3 mg
Acronym: LETHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Geltrude Mingrone, Principal Investigator, Catholic University of the Sacred Heart
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0002017056
Record Dates: First submitted 2017-10-30; First posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Obesity
Keywords: obesity; sleeve-gastrectomy; liraglutide; Weight-loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Liraglutide

STUDY DESIGN:
Intervention Model Description: lifestyle modification alone, lifestyle modification and Liraglutide 3 mg daily, sleeve gastrectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lifestyle modification (Active Comparator): 1 month of a VLCD with 865 kcal per day followed by a 12 kcal per kg of body weight of a high-protein, high fat diet for 11 months in association with intensive
  Interventions: Other: lifestyle modification
- Lifestyle modification plus Liraglutide 3 mg (Experimental): 1 month of a VLCD with 865 kcal per day followed by a 12 kcal per kg of body weight of a high-protein, high fat diet for 11 months in association with intensive. The patients will also receive Liraglutide 3 mg daily sc.
  Interventions: Drug: LIRAGLUTIDE 3 Mg/0.5 mL (18 Mg/3 mL) SUB-Q PEN INJECTOR (ML); Other: lifestyle modification
- Sleeve Gastrectomy (Active Comparator): The patients will undergo laparoscopic sleeve gastrectomy
  Interventions: Other: sleeve gastrectomy

INTERVENTIONS:
Drug: LIRAGLUTIDE 3 Mg/0.5 mL (18 Mg/3 mL) SUB-Q PEN INJECTOR (ML)
  Arms: Lifestyle modification plus Liraglutide 3 mg
Other: lifestyle modification
  Arms: Lifestyle modification; Lifestyle modification plus Liraglutide 3 mg
Other: sleeve gastrectomy
  Arms: Sleeve Gastrectomy

SUMMARY:
Background/Objectives: Only 1% of the clinically eligible subjects receive surgical treatment for their obesity, thus other options should be investigated. In this study we aim to assess the effect of intensive-lifestyle-modification(ILM) with or without Liraglutide-3mg daily versus sleeve-gastrectomy(SG) on BMI at 1-year.

Subjects/Methods: In this study performed in a University Hospital in Italy, non-diabetic patients eligible for bariatric-surgery are recruited from the weight loss clinic and have the option to choose within three possible weight-loss programs up to complete the allocation of 25 subjects in each arm matched by BMI and age. ILM consists in 600kcal very-low-calorie-diet(VLCD) for 1 month followed by 12kcal/kgbw high-protein, high-fat-diet for 11 months plus 30minutes brisk-walk daily and at least 3 hours aerobic-exercise weekly. SG patients have 1-month VLCD and free-diet thereafter. Patients are evaluated at baseline and at 1,3,6,9 and 12months.

DETAILED DESCRIPTION:
Obesity is associated with major chronic diseases, including type 2 diabetes (T2D) and cardiovascular disease (CVD) 1-3. The number of subjects affected by morbid obesity or class III obesity (BMI≥40 kg/m2) is rapidly increasing 4 and contributed to 20% of the total per capita health-care expenditures in 2000 in the United States 5 .

Subjects with a body mass index (BMI) >40 kg/m2 or >35 kg/m2 in the presence of obesity complications are eligible for bariatric surgery 6 . The mortality rate after bariatric surgery is low, being 0.08% within 30 days and 0.31% after 30 days 7, and bariatric surgery has shown many health benefits including reduction of long term mortality 8 and type 2 diabetes remission (T2D) 9-11., However, due to the perception that bariatric surgery is a risky procedure among the general public and insurance companies or other health care providers only 1% of the clinically eligible subjects receive surgical treatment for their obesity 12.

The largest portion of patients eligible for bariatric surgery but who are not willing to be operated or cannot undergo surgery for other reasons should be offered, however, with other therapeutic options. To this end a pilot study to determine the efficacy of an intensive lifestyle modification (ILM) with or without 3 mg daily Liraglutide versus bariatric surgery with free diet and free physical activity was designed. In the medical arms the patients were also invited to contact the dietitian and the physician every week by email or by phone to assure a tight weight control. The allocation of the patients, all of them eligible for bariatric surgery, was on a voluntary basis, i.e. they were invited to decide their allocation in one of the 3 arms of the study matched by BMI and age.

Liraglutide, a glucagon-like peptide-1 analog, approved for the treatment of obesity at the dose of 3 mg per day and commercialized under the name of Saxenda, was proved to reduce body weight after 56 weeks by 8.4±7.3 kg as compared with a mean of 2.8±6.5 kg in the patients under placebo 13 . Importantly, the weight reduction is maintained up to 3 years as shown by LeRoux et al. 14.

However, this degree of weight loss is generally considered insufficient by patients who would like to be considered for bariatric surgery.

A 12 week VLCD was reported to allow a weight reduction of about 20 kg in men and of near 16 kg in women 15. However, the weight-reducing effect of a VLCD is temporary and must be combined with other methods to maintain the weight loss. Low-carbohydrate, high-fat, high-protein diet is associated with a relevant weight loss and elevated satiating effects as well as with maintenance or accretion of lean body mass 16,17.

In this study it was hypothesized that a VLCD for 1 month might match in the two medical arms the weight loss reached with SG, thus giving more motivation to the patients to continue the diet. The aim of the study is to find other avenues than bariatric surgery to treat obese patients obtaining a relevant weight loss that can satisfy morbidly obese subjects.

Therefore, this trial included a VLCD for the first month in order to match the diet usually prescribed after bariatric surgery and the following diet will be a low-carbohydrate, high-fat, high-protein diet to achieve a substantial weight loss.

Among the surgical procedures sleeve gastrectomy (SG) was chosen since it has increased markedly in the past few years and has earned a place as a primary bariatric surgery 18.

ELIGIBILITY:
Inclusion Criteria:

Age ranging from 18 to 70 years, stable body weight in the previous 6 months body mass index (BMI expressed in kg/m2) >35 if comorbidity (hypertension, sleep apnea, severe hip or knee arthritis) are present or >40 kg/m2.

Exclusion Criteria:

Type 1 or 2 diabetes, previous bariatric surgery, a history of pancreatitis, a history of major depressive or other severe psychiatric disorders, a family or personal history of multiple endocrine cancer type 2 or familial medullary thyroid carcinoma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-04-10 (Actual)

PRIMARY OUTCOMES:
Change of baseline BMI | 1 year
  percent variation of BMI with respect to baseline value

SECONDARY OUTCOMES:
changes of baseline weight plasma | 1 year
  percent variation of variables with respect to baseline value
changes in body composition | 1 year
  percent variation of variables with respect to baseline value
changes in plasma glucose | 1 year
  percent variation of variables with respect to baseline value
changes in HOMA-IR | 1 year
  percent variation of variables with respect to baseline value
changes in blood pressure | 1 year
  percent variation of variables with respect to baseline value
changes in lipid profile | 1 year
  percent variation of variables with respect to baseline value

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University School of Medicine, Rome, Italy